CLINICAL TRIAL: NCT00672555
Title: Prospective Evaluation of Feasibility and Results of the Treatment of Pilonidal Sinus by Excision and Covering of the Defect With a Limberg-flap.
Brief Title: Limberg-flap: Prospective Data Collection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Dr. med. D. Germann; (MD), Cantonal Hospital of St. Gallen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EKSG 07/050/2B
Record Dates: First submitted 2008-05-01; First posted 2008-05-06 (Estimated); Results first posted 2011-06-29 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Pilonidal Sinus
Keywords: pilonidal sinus; recurrence; Limberg flap
MeSH Terms: conditions — Pilonidal Sinus; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pilonidal Sinus T. With Limberg F. (Experimental): All patients treated by excision and covering of the defect by a Limberg-flap, who gave their informed consent to participate in the study, as there is only one study group.
  Interventions: Procedure: Limberg-flap

INTERVENTIONS:
Procedure: Limberg-flap — Complete excision of the pilonidal sinus and covering of the defect by a Limberg-flap from one buttock
  Other Names: Romboid-flap

SUMMARY:
The investigators think, that the treatment of pilonidal sinus with excision and covering of the defect with a Limberg-flap is a very good treatment option. The investigators are introducing this treatment for recurrences of this illness in our clinic and want to analyse the feasibility, the results, the complications and the patients opinion after the treatment.

If the results are good, a prospective randomised study is a further option.

DETAILED DESCRIPTION:
1. Patients, that come to our clinic with problems caused by a pilonidal sinus are informed about the different treatment options of the illness.

   * If the patient suffers of a recurrence of the illness, a complete excision, followed by a covering of the defect with a Limberg-flap is recommended.
   * If the patient has the first time problems by a pilonidal sinus, we recommend an open limited excision of the fistulas.
   * In cases with acute infected situation, we first conduct a very limited incision/excision and treat them with antibiotics. The treatments mentioned before are in such cases offered 3 to 4 Weeks after the fist little operation.
2. All Patients, that wish their pilonidal sinus treated with a complete excision followed by a covering of the defect with a Limberg-flap, are asked if they are willing to participate in the observational study.
3. Patients, who gave their informed consent for the operation and the study are included.
4. Preoperative data are recorded.
5. The patients are operated on and intraoperative data (e.g. how big was the flap) are recorded.
6. After 3 Weeks the patients are checked and complications, happiness and duration of the time off work are recorded.
7. After a year the patients are contacted by sending them a postal questionnaire, which they send back to us. Additionally the are contacted by phone. Recurrence, other complications and their opinion concerning the treatment and its consequences are recorded.

ELIGIBILITY:
Inclusion Criteria:

* Recurrence or persistence of a pilonidal sinus
* Elective Limberg-flap operation
* Written informed consent of the patient for the operation and participation of the study

Exclusion Criteria:

* Doubts of the capability of the patient to understand the study or to decide.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-08; Primary Completion 2009-01 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Marti, M D, Principal Investigator — Department of surgery, Cantonal hospital of St. Gallen; Franc H Hetzer, M D, Study Chair — Department of surgery, Cantonal hospital of St. Gallen
Locations (2):
- Switzerland (2):
  - Department of sugery, Cantonal hospital of St. Gallen, Rorschach, Canton of St. Gallen
  - Department of surgery, Cantonal hospital of St. Gallen, Sankt Gallen, Canton of St. Gallen

REFERENCES:
- [Background] Kapp T, Zadnikar M, Hahnloser D, Soll Ch, Hetzer FH. [New concept in the treatment of the pilonidal sinus]. Praxis (Bern 1994). 2007 Aug 2;96(31-32):1171-6. doi: 10.1024/1661-8157.96.31.1171. German. PMID 17726856
- [Background] Dunker MS, Stiggelbout AM, van Hogezand RA, Ringers J, Griffioen G, Bemelman WA. Cosmesis and body image after laparoscopic-assisted and open ileocolic resection for Crohn's disease. Surg Endosc. 1998 Nov;12(11):1334-40. doi: 10.1007/s004649900851. PMID 9788857
- [Result] Muller K, Marti L, Tarantino I, Jayne DG, Wolff K, Hetzer FH. Prospective analysis of cosmesis, morbidity, and patient satisfaction following Limberg flap for the treatment of sacrococcygeal pilonidal sinus. Dis Colon Rectum. 2011 Apr;54(4):487-94. doi: 10.1007/DCR.0b013e3182051d96. PMID 21383571

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients meeting the inclusion criteria during the study recruiting period, who gave their consent included.
Pre-assignment Details: 1 patient excluded because of mental handicap
Groups:
- Pilonidal Sinus Treated With Limberg Flap: All patients treated by excision and covering of the defect by a Limberg-flap, who gave their informed consent to participate in the study, as there is only one study group.
Period: Overall Study
Arm/Group | Pilonidal Sinus Treated With Limberg Flap
Started | 70
Completed | 64 (All patients were seen at 3 weeks in the outpatient clinic.)
Not Completed | 6
Not completed — Lost to Follow-up | 4
Not completed — Did not want to answer questionnaire | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pilonidal Sinus Treated With Limberg Flap
Number analyzed (Participants) | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 70
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 26.1 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 57
Region of Enrollment [Number; unit: participants]
  Switzerland | 70

OUTCOME MEASURES:

1. Primary Outcome: Recurrence of a Pilonidal Sinus After Operation Using a Limberg-flap Procedure
Description: At 1 year all patients were assessed. Patients with a recurrence of a pilonidal sinus were counted. The result is given as number of patients suffering from a recurrence.
Time Frame: 1 year
Population: Per protocol:
  All patients treated in the study period, who gave their informed consent and meet the inclusion criteria, as well did not have any reason for exclusion were enrolled prospectively
Measure: Number; unit: participants
Arm/Group | Pilonidal Sinus Treated With Limberg Flap
Number analyzed (Participants) | 70
participants | 1

2. Secondary Outcome: Minor Complications (Wound Complications)
Description: All wound complications were assessed; part of them being only very minor dehiscences or slight infections. They were assessed in the outpatients clinic at 3 Weeks and in the follow-up control initiated at 1 year. All patients suffering from a wound complication that occurred in the first year were counted.
Time Frame: 1 year
Measure: Number; unit: participants
Arm/Group | Pilonidal Sinus Treated With Limberg Flap
Number analyzed (Participants) | 70
participants | 18

3. Secondary Outcome: Reoperations Needed for Treatment of Complication
Description: All patients were seen at the outpatients clinic at 3 weeks. Follow-up control was initiated at 1 year.
  All reoperations that were done were assessed and measured.
Time Frame: 1year
Measure: Number; unit: Reoperations
Arm/Group | Pilonidal Sinus Treated With Limberg Flap
Number analyzed (Participants) | 70
Reoperations | 6

4. Secondary Outcome: Patient Overall Satisfaction With Procedure
Description: Follow-up was initiated at 1 year. A postal questionnaire was sent to the patients with a VAS assessing overall satisfaction. Possible values were: lowest: 0; highest 10.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pilonidal Sinus Treated With Limberg Flap
Number analyzed (Participants) | 70
Units on a scale | 7.6 (2.3)

5. Secondary Outcome: Body Image Score
Description: Patients was sent a postal questionnaire at 1 year, assessing body image with the body image questionnaire adapted from Dunker et al. Body image score resulting form 5 questions: worst 5; best 20.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pilonidal Sinus Treated With Limberg Flap
Number analyzed (Participants) | 70
Units on a scale | 17.9 (2.6)

6. Secondary Outcome: Cosmetic Score
Description: Patients was sent a postal questionnaire at 1 year, assessing cosmesis with the body image questionnaire adapted from Dunker et al. Cosmetic score resulting form 3 questions: worst 3; best 24.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pilonidal Sinus Treated With Limberg Flap
Number analyzed (Participants) | 70
Units on a scale | 16.4 (4.3)

ADVERSE EVENTS:
Time Frame: 1 years
Arm/Group | Pilonidal Sinus Treated With Limberg Flap
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 18/70
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pilonidal Sinus Treated With Limberg Flap (N=70)
Complication (Infections and infestations) | 18 (18) — All complications were assessed. Apart from a bleeding which stopped with compression, all were infections or wound dehiscences.

LIMITATIONS AND CAVEATS:
Study was conducted as planned. A long time was needed to get the follow-up information.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes